CLINICAL TRIAL: NCT04021485
Title: 5-year Follow-up of the BETADOSE Trial: Non-inferiority of a 50% Dose Reduction of Antenatal Betamethasone Therapy on the Neurodevelopment of Children Born Before 32 Weeks of Gestation.
Brief Title: BETAmethasone Dose Reduction: Non-Inferiority on the Neurocognitive Outcomes of Children Born Before 32 Weeks of Gestation
Acronym: BETANINO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: K170920J
Record Dates: First submitted 2019-07-08; First posted 2019-07-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Premature Childbirth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neurodevelopmental assessment (Other): As part of the usual follow-up of premature children, a follow-up consultation is planned around the age of 5 years. During this visit, a neurodevelopmental assessment will be carried out for the Betanino study. The duration of this evaluation is evaluated around 3h in total.
  Interventions will include:
  * Standardized neurological exam
  * Morphometric measurements including height, weight, head circumference
  * Blood pressure measurement
  * Multiple aspects of cognition using ancillary indexes of WPPSI-IV subtests, NEPSY-II subtests,
  * Social Relativeness, using Social Relativeness Scale parental questionnaire,
  * Parental stress using PSI questionnaire
  Interventions: Other: neurodevelopmental assessment

INTERVENTIONS:
Other: neurodevelopmental assessment — As part of the usual follow-up of premature children, a follow-up consultation is planned around the age of 5 years. During this visit, a neurodevelopmental assessment will be carried out for the Betanino study. The duration of this evaluation is evaluated around 3h in total.
  Interventions will include:
  * Standardized neurological exam
  * Morphometric measurements including height, weight, head circumference
  * Blood pressure measurement
  * Multiple aspects of cognition using ancillary indexes of WPPSI-IV subtests, NEPSY-II subtests,
  * Social Relativeness, using Social Relativeness Scale parental questionnaire,
  * Parental stress using PSI questionnaire

SUMMARY:
Maternal antenatal corticosteroid therapy is the last major advance in the antenatal management of fetuses to prevent neonatal complications associated with prematurity. Long-term neurological outcomes in infants exposed to antenatal steroids have been assessed in few cohorts and suggest that this therapy is able to prevent some neurodevelopmental impairments including cerebral palsy. While >85% of neonates born very preterm in Europe have been exposed to antenatal betamethasone, Cochrane collaborative networks stated that trials of dosages comparing different regimens of commonly used corticosteroids are most urgently needed to avoid useless fetal exposure to excessive dosage of corticosteroids.

* Because a half dosage was associated with maximal benefits on lung function in ewes, a randomized controlled trial (BETADOSE, NCT02897076) has been conducted to demonstrate that a 50% reduced betamethasone dose regimen is not inferior to a full dose to prevent respiratory distress syndrome in preterm neonates. BETADOSE trial demonstrated that half dose did not show noninferiority to full antenatal betamethasone dose regimen to prevent severe RDS in preterm neonates while other prematurity-associated complications, including those usually prevented by ACS, did not differ between the two groups.
* Results of the 5-year BETANINO follow-up study of the BETADOSE neonates are needed before deciding whether reducing ACS dose is possible The main hypothesis of BETANINO is that half dose regimen of betamethasone is not inferior to full dose regimen of betamethasone to prevent neurodevelopmental impairments in these high-risk children born very preterm at 5 years of age.

DETAILED DESCRIPTION:
Maternal antenatal corticosteroids (ACS) therapy is considered to be the last major advance in the antenatal management of fetuses at risk of preterm birth. It was adopted worldwide to prevent neonatal death and neonatal complications following preterm birth, including respiratory distress syndrome, necrotizing enterocolitis and severe intraventricular hemorrhage. While short-term benefits of ACS were extensively investigated, long-term neurological outcomes in infants exposed antenatally to betamethasone have been assessed in few cohorts only. A recent report from the Cochrane collaborative network suggest that ACS is able to prevent some neurodevelopmental impairments associated with preterm delivery and related to postnatal adverse events .

As of today, in Europe and France, more than 85% of neonates born very preterm have been exposed to antenatal corticosteroids, mostly betamethasone for a total dose of 24 mg. Cochrane collaborative networks stated that trials of dosages comparing different regimens of commonly used corticosteroids are most urgently needed. Because a half dosage was associated with maximal benefits on lung function in ewes, a randomized controlled trial (BETADOSE, NCT02897076) is currently conducted to demonstrate that a 50% reduced betamethasone dose regimen is not inferior to a full dose regimen to prevent respiratory distress syndrome in neonates. Whatever the results of this ongoing clinical trial, follow-up of infants born from enrolled women is mandatory both to confirm the non-inferiority of the dose reduction on neurocognition and to assess the long-term effect of dose reduction on survival, on complex aspects of cognition, on behavioral aspects and on others neurodevelopmental impairments. Indeed, changes in clinical practices following BETADOSE trials will be depending on both short- and long-term outcomes. If non inferiority is demonstrated, dramatic changes will occur in the clinical use of antenatal betamethasone in women at risk of preterm birth in France and worldwide. If non inferiority is rejected, the neurocognitive follow-up of enrolled patients will be also of interest to (i) assess the long-term impact of the early consequences associated with betamethasone dose reduction and (ii) to find out domains of neurocognitive development sensitive to ACS exposure.

BETANINO study aims at assessing the impact of a 50% dose reduction on neurocognition at 5 years of age in infants born from mothers enrolled in the BETADOSE trial before 32 weeks of gestation, children that are at highest risk of neurocognitive impairments during childhood.

The main hypothesis of this cohort study following a randomized clinical trial is that half dose betamethasone (12 mg) is not inferior to full dose betamethasone (24 mg) to prevent neurodevelopmental impairment in children born very preterm.

ELIGIBILITY:
Inclusion Criteria:

* Singleton child born from mother enrolled in the BETADOSE trial,
* Gestational age at birth less than 32 weeks of gestation,
* Age ≥ 5 years and < 6 years, alive and not lost of follow up
* Informed consent of the holder (s) of the exercise of parental authority
* Affiliation to a social security scheme.

Exclusion Criteria:

* Major malformations and chromosomal aberrations evidenced after birth,
* Parents' refuse to participate.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 643 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
neurocognitive development | 5 years
  Cognition will be assessed by certified neuropsychologists at 5 years of age using full scale IQ generated by Wechsler Preschool and Primary Scale of Intelligence (WPPSI-IV) test.

SECONDARY OUTCOMES:
5-year survival without moderate-to-severe impairment | 5 years
neurocognitive development | 5 years
  Measured by WPPSI-IV subtests
Parental stress | 5 years
  Using Social Relativeness Scale
Parental stress | 5 years
  Parental stress using PSI questionnaire All assessments will be based on internationally recognized tests that have been validated for infants at 3 years of age and conducted by certified neuropsychologists.
cerebral palsy | 5 years
  cerebral palsy using the GMFCS notation system,
neurocognitive development | 5 years
  Measured by NEPSY subtests

CONTACTS AND LOCATIONS:
Overall Officials: Biran Valerie, PHD, Principal Investigator — APHP; Baud Olivier, PHD, Study Chair — Hôpitaux Universitaires de Genève - Inserm U1141 Hôpital Robert Debré; Schmitz Thomas, PHD, Study Chair — APHP
Locations (1):
- Hôpital Robert Debré, Paris, Pa, France